CLINICAL TRIAL: NCT07333976
Title: o A Prospective, Randomized, Open-Label, Phase II Study Evaluating the Efficacy of Tadalafil for the Prevention of Docetaxel-Induced Peripheral Neuropathy in Patients With Metastatic Prostate Cancer
Brief Title: o Tadalafil for Prevention of Docetaxel-Induced Peripheral Neuropathy in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, MING-HSIN, YANG, DR., Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2-107-05-167DIPN
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Metastatic Disease; Chemotherapy Induced Peripheral Neuropathy (CIPN); Neurotoxicity
Keywords: tadalafil; docetaxel; Peripheral Neuropathy; Supportive Care; Prevention
MeSH Terms: conditions — Neurotoxicity Syndromes; Peripheral Nervous System Diseases | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil Group (Experimental) (Experimental): Patients receive Docetaxel chemotherapy plus Tadalafil.
  Interventions: Drug: Tadalafil 5 mg
- Control Group (No Intervention) (No Intervention): Patients receive Docetaxel chemotherapy with standard supportive care alone.

INTERVENTIONS:
Drug: Tadalafil 5 mg — 5 mg administered orally on alternate days (every 48 hours), starting from the first day of chemotherapy cycle 1 until the completion of chemotherapy.
  Arms: Tadalafil Group (Experimental)

SUMMARY:
Docetaxel is a standard chemotherapy for metastatic prostate cancer but is associated with dose-limiting peripheral neuropathy. Currently, no pharmacologic agents are established for prevention. Tadalafil, a PDE5 inhibitor, may improve microvascular perfusion and offer neuroprotection. This randomized phase II trial evaluates whether concurrent use of tadalafil (5 mg every 2 days) reduces the incidence and severity of docetaxel-induced peripheral neuropathy compared to standard care in patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma.
* Metastatic hormone-sensitive (mHSPC) or castration-resistant prostate cancer (mCRPC).
* Scheduled to receive docetaxel chemotherapy (50 mg/m^2 biweekly).
* ECOG performance status 0-2.
* Adequate bone marrow, hepatic, and renal function.

Exclusion Criteria:

* Pre-existing peripheral neuropathy (CTCAE grade >= 1).
* Prior treatment with taxane-based chemotherapy.
* Concurrent use of nitrates or nitric oxide donors.
* Severe cardiovascular disease (e.g., unstable angina, recent myocardial infarction within 6 months).
* Known hypersensitivity to tadalafil or PDE5 inhibitors.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Peripheral Neuropathy | From baseline up to the completion of 6 cycles of chemotherapy (approximately 12 weeks).
  Defined as the proportion of patients developing sensory neuropathy Grade > 1 according to NCI-CTCAE version 5.0 criteria.

SECONDARY OUTCOMES:
Incidence of Moderate to Severe Neuropathy | Up to 12 weeks.
  Proportion of patients developing CTCAE Grade > 2 sensory neuropathy (limiting instrumental activities of daily living).
Patient-Reported Neuropathy Symptoms (EORTC QLQ-CIPN20) | Assessed at baseline and before each chemotherapy cycle (every 2 weeks) up to 12 weeks.
  Change from baseline in sensory and motor scores assessed by the EORTC QLQ-CIPN20 questionnaire. Scores range from 0 to 100, with higher scores indicating worse symptoms.
Oncological Efficacy (PSA Response) | Up to 12 weeks.
  Percentage change in Prostate-Specific Antigen (PSA) levels from baseline to the end of treatment. This is a safety endpoint to ensure non-inferiority.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: No